CLINICAL TRIAL: NCT04005560
Title: Patient's Quality of Life Assessment 5 to 10 Years After Hospitalization in Intensive Care Unit for a Severe Bacterial Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC19_0128
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Quality of Life; Sequela
Keywords: severe bacterial infection; quality of life; long term sequela; pediatric intensive care unit; children
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Other): Score of PedSQL who is the Pediatric Quality of Life Questionnaire
  Interventions: Other: no interventional study

INTERVENTIONS:
Other: no interventional study — no interventional study

SUMMARY:
The aim of this study is to assess patient's quality of life 5 to 10 years after a severe bacterial infection with hospitalization in a intensive unit care. The population is derived from the DIABACT III study. The investigators will include every patient still alive. To evaluate our question, patients and their parents will answer quality of life questionnaires. The investigators will also have telephone interviews with the parents to know somatic and psychological effects on their child.

The investigators will see if quality of life and sequelae differ depending on various studied factors.

DETAILED DESCRIPTION:
The aim of this study is to assess patient's quality of life 5 to 10 years after hospitalization in intensive car unit for a severe bacterial infection. The population is derived from DIABACT III study, and includes all patients still alive.

To evaluate their quality of life, patients and parents will answer specific questionnaries. The Pediatric Quality of Life inventory (PedSQL) has various versions for children depending on their age, adults and parents. The investigators will get physical, emotional, social and academic scores.

To assess somatic and psychological effect after the severe bacterial infection, the investigators will have telephone interviews with the parents, with many questions about organs disorders, specialized medical follow-up, medication, need physical or material assistance, financial and psychological family impact… The investigators will examine data from DIABACT III study to assess determinants of the quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Every patients from DIABACT III study still alive at the beginning of this study

Exclusion Criteria:

* Patients who did not respond to the questionnaire
* Inability to contact the patient and family
* No fixed postal address

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
This quality of life will be evaluated by a questionnaire, the Pediatric Quality of Life inventory. | 6 months
  The Pediatric Quality of Life inventory questionnaire has various versions depending on the patient age, from 5 years old to adult age. Patients will answers many questions in the academic, emotional, physical and social fields. It exists the same questionnaire adapted for parents. At the end, there is a score for each field and a total score.

SECONDARY OUTCOMES:
Identify quality of life determinants. | 6 months
  DIABACT III database has factors that could affect quality of life.
Assess long-term sequelae: evaluate somatic and psychological effects. We will have telephone interviews with the parents. | 6 months
  During the telephone interview, we will ask many questions about organs disorders and psychological disorders (Strenghts and Difficulties Questionnaire), specialized medical follow-up, medication, need physical or material assistance, financial and psychological family impact

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided